CLINICAL TRIAL: NCT06857474
Title: The Effect of Bristle Brush, Rubber Cup, and Air Polishing on Tooth Surface Roughness of Scaled Teeth: A Randomized Controlled Trial Study Using Scanning Electron Microscope: Randomized Controlled Trial
Brief Title: The Effect of Bristle Brush, Rubber Cup, and Air Polishing on Tooth Surface Roughness of Scaled Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: Khyber College of Dentistry (KCD) Peshawar (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2024/014
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Periodontal Diseases; Tooth Abrasion; Dental Plaque
Keywords: Tooth roughness; Dental polishing; Bristal Brush; Periodontology
MeSH Terms: conditions — Periodontal Diseases; Tooth Abrasion; Dental Plaque

STUDY DESIGN:
Intervention Model Description: The study compares the effects of three different polishing methods (bristle brush, rubber cup, and air polishing) on tooth surface roughness in a randomized controlled trial with a control group.
Who Masked: Participant, Care Provider
Masking Description: This study follows a double-blind approach where both the SEM technician capturing micrographs and the analyst evaluating surface roughness will be blinded to the specific group allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bristle Brush Polishing Group (Experimental): After ultrasonic scaling, teeth will be polished using a bristle brush attached to a low-speed contra-angle handpiece with prophylaxis paste in a circular motion for 10 seconds.
  Interventions: Procedure: Bristle Brush Polishing
- Rubber Cup Polishing Group (Experimental): After ultrasonic scaling, teeth will be polished using a rubber cup attached to a low-speed contra-angle handpiece with prophylaxis paste in a circular motion for 10 seconds.
  Interventions: Procedure: Rubber Cup Polishing
- Air Polishing Group (Experimental): After ultrasonic scaling, teeth will be polished using sodium bicarbonate air polishing with an air polishing device in a circular motion for 10 seconds.
  Interventions: Procedure: Air Polishing
- Control Group (Active Comparator): Teeth in this group will undergo ultrasonic scaling only, with no additional polishing procedures.
  Interventions: Procedure: Ultrasonic Scaling

INTERVENTIONS:
Procedure: Bristle Brush Polishing — After ultrasonic scaling, teeth will be polished using a bristle brush attached to a low-speed contra-angle handpiece with prophylaxis paste in a circular motion for 10 seconds.
  Arms: Bristle Brush Polishing Group
Procedure: Rubber Cup Polishing — After ultrasonic scaling, teeth will be polished using a rubber cup attached to a low-speed contra-angle handpiece with prophylaxis paste in a circular motion for 10 seconds.
  Arms: Rubber Cup Polishing Group
Procedure: Air Polishing — After ultrasonic scaling, teeth will be polished using sodium bicarbonate air polishing with an air polishing device in a circular motion for 10 seconds.
  Arms: Air Polishing Group
Procedure: Ultrasonic Scaling — Teeth in the control group will undergo ultrasonic scaling only, with no additional polishing procedures.
  Arms: Control Group

SUMMARY:
This study investigates the effects of three polishing methods using a bristle brush, rubber cup, and air polishing on the surface roughness of scaled human teeth. The study aims to determine which polishing method is most effective in minimizing roughness and preventing plaque accumulation, thus contributing to improved oral health practices.

DETAILED DESCRIPTION:
Tooth surface roughness influences plaque retention and periodontal health. Polishing after scaling helps smoothen enamel surfaces, reducing bacterial adhesion. While various studies have assessed polishing techniques, there are inconsistencies in findings, particularly regarding air polishing vs. rubber cup polishing. Additionally, most studies focus on bovine teeth or indirect restorative materials rather than extracted human teeth. Using a randomized controlled trial (RCT) design, 56 extracted teeth will be divided into four groups: a control group (no polishing) and three experimental groups subjected to different polishing techniques. Surface roughness will be analyzed using a Scanning Electron Microscope (SEM). This study aims to fill these research gaps and provide region-specific data by determining which polishing method is most effective in minimizing roughness and preventing plaque accumulation, thus contributing to improved oral health practices.

ELIGIBILITY:
Inclusion Criteria:

* Extracted human teeth with intact buccal or lingual surfaces.
* Patients with a history of trauma affecting the oral cavity will be eligible, provided they meet other criteria (e.g., intact buccal or lingual surfaces).
* Male and female patients aged 18 years and above.

Exclusion Criteria:

* Teeth with restorations, caries, fractures, or significant developmental defects (e.g., amelogenesis imperfecta, dentinogenesis imperfecta , fluorosis etc).
* Patients with systemic disease such as diabetes mellitus, cardiovascular disorders or any other condition will be excluded.
* Mentally impaired patient.
* Patients who have undergone scaling and polishing within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-28 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Tooth Surface Roughness | Immediately after intervention (post-polishing SEM analysis).
  The arithmetic mean roughness (Ra) and root mean square roughness (Rq) of the enamel surface will be measured using Scanning Electron Microscopy (SEM) analysis and ImageJ software. This will assess the effectiveness of different polishing techniques in reducing surface roughness after ultrasonic scaling.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Khan, BDS, Principal Investigator — Khyber College of Dentistry, Peshawar; Syed Muaz Masoom Shah, BDS,MDS,PHD, Principal Investigator — Khyber College of Dentistry, Peshawar; Mehwish Rasool, BDS, Principal Investigator — Khyber College of Dentistry, Peshawar; Syed Muhammad Shabbir Ali Naqvi, PhD*, Principal Investigator — Khyber Medical University Peshawar
Locations (1):
- Khyber College of Dentistry, Peshawar, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The study will share de-identified individual participant data (IPD), including surface roughness measurements obtained from Scanning Electron Microscopy (SEM) analysis, as well as statistical findings related to different polishing techniques. The shared dataset will help researchers conduct secondary analyses and compare results with similar studies.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be made available 6 months after the study's completion and will remain accessible for a period of 5 years to facilitate further research.
Access Criteria: Access to the data will be granted to qualified researchers upon submission of a formal request that includes a research proposal outlining the intended use of the data. Requests will be reviewed by the study investigators and ethical review committee to ensure compliance with data privacy regulations.

REFERENCES:
- [Background] Al-Amri I, Albounni R, Binalrimal S. Evaluation of the effect of soft drinks on the surface roughness of dental enamel in natural human teeth. F1000Res. 2021 Nov 10;10:1138. doi: 10.12688/f1000research.55556.1. eCollection 2021. PMID 35186274
- [Background] Mohabatpour F, Chen X, Papagerakis S, Papagerakis P. Novel trends, challenges and new perspectives for enamel repair and regeneration to treat dental defects. Biomater Sci. 2022 Jun 14;10(12):3062-3087. doi: 10.1039/d2bm00072e. PMID 35543379
- [Background] Jakubovics NS, Goodman SD, Mashburn-Warren L, Stafford GP, Cieplik F. The dental plaque biofilm matrix. Periodontol 2000. 2021 Jun;86(1):32-56. doi: 10.1111/prd.12361. Epub 2021 Mar 10. PMID 33690911
- [Background] Wei Y, Dang GP, Ren ZY, Wan MC, Wang CY, Li HB, Zhang T, Tay FR, Niu LN. Recent advances in the pathogenesis and prevention strategies of dental calculus. NPJ Biofilms Microbiomes. 2024 Jul 13;10(1):56. doi: 10.1038/s41522-024-00529-1. PMID 39003275
- [Background] Chowdhary Z, Mohan R. Efficiency of three different polishing methods on enamel and cementum: A scanning electron microscope study. J Indian Soc Periodontol. 2018 Jan-Feb;22(1):18-24. doi: 10.4103/jisp.jisp_40_17. PMID 29568167